CLINICAL TRIAL: NCT01779219
Title: The Safety and Effectiveness of Low Field Intraoperative MRI-guidance in Frameless Stereotactic Biopsies of Brain Tumours - a Prospective Randomized Trial
Brief Title: Intraoperative MRI-guidance in Frameless Stereotactic Biopsies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator has changed his employee and the country of residence.
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Marcin Czyz, M.D., Ph.D., Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STAT2009
Record Dates: First submitted 2013-01-15; First posted 2013-01-30 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Primary Brain Tumour
Keywords: intraoperative magnetic resonance; stereotactic biopsy; brain tumor; frameless stereotaxy; image-guided neurosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Neuronavigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iMRI-guided (Active Comparator): Intervention: iMRI-guided brain tumour biopsy. The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a 0.15-T constant magnet imager will be used in all cases. After the patient's positioning, the preoperative reference examination is routinely carried out. The entry point, target and optimal biopsy trajectory are then defined by the operator on the basis of the obtained iMRI images. Serial tissue samples are collected. Following each operation, a control iMRI (T1-weighted, axial, 4 mm scan examination) is routinely performed to confirm and document the proper targeting and to exclude postoperative hyperacute intraparenchymal bleeding.
  Interventions: Device: iMRI-guided brain tumour biopsy
- non-iMRI (Active Comparator): Intervention: Stereotactic frameless brain tumour biopsy. A frameless STx biopsy is performed for each patient from the control group with the use of a neuronavigation system. The entry point, target and optimal biopsy trajectory are defined by the operator before the operation on the basis of the preoperatively obtained high-field MR images with the use of a neuronavigation workstation (Cranial 5, StealthStation Application Software, Medtronic Navigation, Louisville, CO, USA).
  Interventions: Device: Stereotactic frameless brain tumour biopsy

INTERVENTIONS:
Device: iMRI-guided brain tumour biopsy — The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a 0.15-T constant magnet was used in all procedures.
  Other Names: iMRI
  Arms: iMRI-guided
Device: Stereotactic frameless brain tumour biopsy — The entry point, target and optimal biopsy trajectory were defined by the operator before the operation on the basis of the preoperatively obtained high-field MR images with the use of a neuronavigation workstation (Cranial 5, StealthStation Application Software, Medtronic Navigation, Louisville, CO, USA).
  Other Names: Neuronavigation; Non-iMRI
  Arms: non-iMRI

SUMMARY:
Background: The aim of the study was to assess the safety and effectiveness of stereotactic brain tumour biopsy (STx biopsy) guided by low-field intraoperative MRI (iMRI) in comparison with its frameless classic analogue based on a prospective randomized trial.

Patients are prospectively randomized into a low-field iMRI group and a control group that undergo a frameless STx biopsy. The primary endpoints of the analysis are: postoperative complication rate and diagnostic yield, and the secondary endpoints: length of hospital stay and duration of operation.

DETAILED DESCRIPTION:
INTRODUCTION Stereotactic brain biopsy (STx biopsy) offers a relatively straightforward, accurate and safe method of obtaining diagnostic tissue. Frameless computer-based neuronavigation is now widely used in brain tumor surgery. It has many advantages over frame-based techniques and provides similar accuracy to the rigid frame. One of the methods applied to improve diagnostic yield and safety is the usage of intraoperative magnetic resonance imaging (iMRI), proposed by Bernays et al. in 2002.

Besides the obvious indications given in previous papers, including STx biopsy of very small, deeply localized or cystic lesions, iMRI guidance is particularly useful in two cases. The first one is when a satisfactory 3D volume modality cannot be obtained during preoperative high-field diagnostic MR imaging. When using iMRI there is no need to perform preoperative 3D imaging of any kind and manually register the patient's head in a neuronavigation system before the operation, which helps to significantly improve the workflow. In our study the total amount of patients with insufficient neuroimaging - admitted from outside medical centers - is over 30%. The second case is for teaching purposes - frameless iMRI guided STx biopsy, is relatively uncomplicated and technically straightforward and can be introduced as the first procedure during training in neurosurgical intraoperative imaging.

Although the usefulness of ultra-low-field iMRI in STx biopsy was subsequently confirmed by other authors, according to our knowledge no previous published studies have compared iMRI to preoperative MRI for brain tumor biopsy according to evidence-based medicine guidelines (EBM). Though this method has been subject to slight criticism, it has been consequently applied in neurosurgical daily practice in recent years.

The aim of our study was to verify the safety and effectiveness of the STx biopsy guided by low-field iMRI in comparison with its frameless classic analogue basing on a prospective randomized parallel-group, controlled trial. In the current paper we present the study design and results of the interim analysis.

MATERIAL AND METHODS

Patients Patients who are - following contemporary recommendations - scheduled to undergo STx biopsy, are prospectively recruited for the study. Each patient sign a written consent to participate in the study.

Inclusion criteria The inclusion criteria were as follows: male and female patients ≥ 18 years with supratentorial brain tumor scheduled to undergo STx biopsy. The estimated number of patients needed to reveal the difference of over 5% between primary endpoints' - diagnostic yield and complications ratio - at the level of significance 0.05 and power 80% was 465 per each arm.

Exclusion criteria Patients unable to provide informed consent and those with metal implants which could prevent or influence the head MR study were excluded from the study.

Allocation Patients were prospectively allocated by minimization according to demographic (gender, age) and epidemiologic data (preoperative Eastern Cooperative Oncology Group Performance Status-ECOG- a scale providing information about neurological and social status of a patient with oncological disease, maximum tumor diameter, presence of contrast enhancement, independent risk factors of hemorrhage - basal and thalamic localization and preoperative diabetes) into the iMRI and the control group.

Intervention After being transferred to the operating room each patient was sedated with an intravenous infusion of Remifentanil with passive oxygen therapy and monitoring of vital functions. Additionally, the sites of head holder pins and skin incision were anaesthetized with 1% Lignocaine. All biopsies in both groups were performed via a 6 mm burr-hole with the use of the Vertec system (Medtronic Navigation, Louisville, CO, USA). A passively navigated side cut 2.2 mm biopsy needle was used. All operations were performed by one of the three first authors.

In the iMRI-guided group the head of each patient was immobilized with a 3-pin iMRI-compatible head holder. The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a 0.15-T constant magnet was used in all procedures. Subsequently, after the patient's positioning, the preoperative reference examination was routinely carried out (T1+gadolinum, T2 or FLAIR weighted - depending on the pathology, axial 4 mm scans). Images were automatically transferred into the neuronavigation system (StealthStation, Medtronic Navigation, Louisville, CO, USA). The entry point, target and optimal biopsy trajectory were then defined by the operator on the basis of the obtained iMRI images. Serial tissue samples (4 from the central and another 4 from the marginal part of the tumor) were collected according to the modified protocol described by Shooman et al., which made use of intraoperative histopathological examination obsolete. Following each operation, a control iMRI (T1-weighted, axial, 4 mm scan examination) was routinely performed to confirm and document the proper targeting and - as proposed by Bernays et al. - to exclude postoperative hyperacute intraparenchymal bleeding.

A frameless STx biopsy was performed for each patient from the control group with the use of a neuronavigation system. The entry point, target and optimal biopsy trajectory were defined by the operator before the operation on the basis of the preoperatively obtained high-field MR images with the use of a neuronavigation workstation (Cranial 5, StealthStation Application Software, Medtronic Navigation, Louisville, CO, USA). Following surgery the specimens were sent for independent histopathological analysis.

Postoperative care Postoperative care was conducted according to standard protocols and clinical guidelines. A postoperative follow-up head CT was subsequently performed 4 to 6 hours after each procedure. All patients were followed up with a clinical examination 2 weeks postoperatively performed by an independent and blinded for the allocation investigator.

Data collection Demographic and epidemiological data were collected prospectively. The primary endpoints were: the ratio of acute postoperative complications and the diagnostic yield. The presence of acute postoperative complication was noted if any of following findings was noted: (wound site infection up to two weeks after the operation, a new neurological deficit developed up to 24 hours following the operation and present in a follow up clinical examination 2 weeks postoperatively), intraparenchymal hematoma with radiological or clinical signs of the intracranial expansion.) and the diagnostic yield. The diagnostic yield was expressed according to the literature as a percentage of patients in whom the histopathological diagnosis was possible on the basis of the biological material obtained during the operation. Secondary endpoints included: the preoperative (LOSpre), postoperative (LOSpost) and total length of hospital stay (LOS) as well as the preparation (Tprep), operation (Top) and total operating room (TOR) time. The LOS and T were routinely measured and recorded in the central hospital files by the independent staff.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients ≥ 18 years
* supratentorial brain tumour
* scheduled to undergo STx biopsy

Exclusion Criteria:

* patients unable to provide informed consent
* metal implants which could prevent or influence the head MR study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wlodzimierz Jarmundowicz, Professor, Study Chair — Wroclaw Medical University
Locations (1):
- Department of Neurosurgery, Wroclaw Medical University, Wroclaw, Poland

REFERENCES:
- [Background] Shooman D, Belli A, Grundy PL. Image-guided frameless stereotactic biopsy without intraoperative neuropathological examination. J Neurosurg. 2010 Aug;113(2):170-8. doi: 10.3171/2009.12.JNS09573. PMID 20136389
- [Background] Czyz M, Tabakow P, Jarmundowicz W, Lechowicz-Glogowska B. Intraoperative magnetic resonance-guided frameless stereotactic biopsies - initial clinical experience. Neurol Neurochir Pol. 2012 Mar-Apr;46(2):157-60. doi: 10.5114/ninp.2012.28258. PMID 22581597
- [Background] Bernays RL, Kollias SS, Khan N, Brandner S, Meier S, Yonekawa Y. Histological yield, complications, and technological considerations in 114 consecutive frameless stereotactic biopsy procedures aided by open intraoperative magnetic resonance imaging. J Neurosurg. 2002 Aug;97(2):354-62. doi: 10.3171/jns.2002.97.2.0354. PMID 12186464
- [Background] Weaver CS, Leonardi-Bee J, Bath-Hextall FJ, Bath PM. Sample size calculations in acute stroke trials: a systematic review of their reporting, characteristics, and relationship with outcome. Stroke. 2004 May;35(5):1216-24. doi: 10.1161/01.STR.0000125010.70652.93. Epub 2004 Mar 18. PMID 15031455
- [Background] Frati A, Pichierri A, Bastianello S, Raco A, Santoro A, Esposito V, Giangaspero F, Salvati M. Frameless stereotactic cerebral biopsy: our experience in 296 cases. Stereotact Funct Neurosurg. 2011;89(4):234-45. doi: 10.1159/000325704. Epub 2011 Jul 21. PMID 21778794
- [Background] Han B, Enas NH, McEntegart D. Randomization by minimization for unbalanced treatment allocation. Stat Med. 2009 Nov 30;28(27):3329-46. doi: 10.1002/sim.3710. PMID 19739238
- [Background] Isaacs D, Fitzgerald D. Seven alternatives to evidence based medicine. BMJ. 1999 Dec 18-25;319(7225):1618. doi: 10.1136/bmj.319.7225.1618. No abstract available. PMID 10600968
- [Background] Kundt G. Comparative evaluation of balancing properties of stratified randomization procedures. Methods Inf Med. 2009;48(2):129-34. doi: 10.3414/ME0538. Epub 2009 Feb 18. PMID 19283309
- [Background] Langen HJ, Kugel H, Ortmann M, Noack M, de Rochemont RM, Landwehr P. [Functional capacity of MRI-compatible biopsy needles in comparison with ferromagnetic biopsy needles. In vitro studies]. Rofo. 2001 Jul;173(7):658-62. doi: 10.1055/s-2001-15844. German. PMID 11512240
- [Background] McGirt MJ, Woodworth GF, Coon AL, Frazier JM, Amundson E, Garonzik I, Olivi A, Weingart JD. Independent predictors of morbidity after image-guided stereotactic brain biopsy: a risk assessment of 270 cases. J Neurosurg. 2005 May;102(5):897-901. doi: 10.3171/jns.2005.102.5.0897. PMID 15926716
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Schulder M, Spiro D. Intraoperative MRI for stereotactic biopsy. Acta Neurochir Suppl. 2011;109:81-7. doi: 10.1007/978-3-211-99651-5_13. PMID 20960325
- [Background] Senft C, Bink A, Franz K, Vatter H, Gasser T, Seifert V. Intraoperative MRI guidance and extent of resection in glioma surgery: a randomised, controlled trial. Lancet Oncol. 2011 Oct;12(11):997-1003. doi: 10.1016/S1470-2045(11)70196-6. Epub 2011 Aug 23. PMID 21868284

RESULTS

PARTICIPANT FLOW:
Groups:
- iMRI: The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a 0.15-T constant magnet is used in all procedures. Subsequently, after the patient's positioning, the preoperative reference examination is routinely carried out (T1+gadolinum, T2 or FLAIR weighted - depending on the pathology, axial 4 mm scans). The entry point, target and optimal biopsy trajectory are then defined by the operator on the basis of the obtained iMRI images. Serial tissue samples (4 from the central and another 4 from the marginal part of the tumour) are collected. Following each operation, a control iMRI (T1-weighted, axial, 4 mm scan examination) is routinely performed to confirm and document the proper targeting and to exclude postoperative hyperacute intraparenchymal bleeding.
  Stereotactic intraoperative magnetic resonance (iMRI)-guided frameless brain tumour biopsy: The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) was used in all cases.
- Non-iMRI: A frameless STx biopsy is performed for each patient from the control group with the use of a neuronavigation system. The entry point, target and optimal biopsy trajectory are defined by the operator before the operation on the basis of the preoperatively obtained high-field MR images with the use of a neuronavigation workstation (Cranial 5, StealthStation Application Software, Medtronic Navigation, Louisville, CO, USA).
  Stereotactic frameless brain tumour biopsy: The entry point, target and optimal biopsy trajectory were defined by the operator before the operation on the basis of the preoperatively obtained high-field MR images with the use of a neuronavigation workstation (Cranial 5, StealthStation Application Software, Medtronic Navigation, Louisville, CO, USA).
Period: Overall Study
Arm/Group | iMRI | Non-iMRI
Started | 21 (First interim analysis) | 21 (First interim analysis)
Completed | 21 (First interim analysis) | 21 (First interim analysis)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- iMRI: The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a 0.15-T constant magnet is used in all procedures. Subsequently, after the patient's positioning, the preoperative reference examination is routinely carried out (T1+gadolinum, T2 or FLAIR weighted - depending on the pathology, axial 4 mm scans). The entry point, target and optimal biopsy trajectory are then defined by the operator on the basis of the obtained iMRI images. Serial tissue samples (4 from the central and another 4 from the marginal part of the tumour) are collected. Following each operation, a control iMRI (T1-weighted, axial, 4 mm scan examination) is routinely performed to confirm and document the proper targeting and to exclude postoperative hyperacute intraparenchymal bleeding.
  Stereotactic intraoperative magnetic resonance (iMRI)-guided frameless brain tumour biopsy: The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with was used in all procedures.
- Total: Total of all reporting groups
Arm/Group | iMRI | Non-iMRI | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (17) | 55 (15) | 54 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  Poland | 21 | 21 | 42
ECOG Performance Status [Median (Inter-Quartile Range); unit: units on a scale] — The ECOG Scale of Performance Status:
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. - Dead
  units on a scale | 2 [1 to 3] | 2 [1 to 2] | 2 [0 to 4]
Maximum tumour diameter [Mean (Standard Deviation); unit: mm] | 48 (19) | 54 (18) | 51 (18)
Tumour enhancement [Number; unit: participants] — Number of participants with contrast-enhancing tumors.
  participants
    Enhancement noted | 16 | 13 | 29
    No enhancement noted | 5 | 8 | 13
Basal localization [Number; unit: participants] — Number of participants with basal localisation of the tumor.
  participants
    basal localisation of the tumor | 7 | 9 | 16
    non-basal localisation of the tumor | 14 | 12 | 26
Thalamic localization [Number; unit: participants] — Number of participants with thalamic localisation of the tumor.
  participants
    thalamic localisation of the tumor | 2 | 4 | 6
    extra-thalamic localisation of the tumor | 19 | 17 | 36
Diabetes [Number; unit: participants] — Number of participants with preoperative diabetes.
  participants
    Diabetes recorded | 6 | 6 | 12
    Diabetes not recorded | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Presenting With Complications
Description: The presence of acute postoperative complication is noted if any of following findings is present: wound site infection up to two weeks after the operation, a new neurological deficit developed up to 24 hours following the operation and present in a follow up clinical examination 2 weeks postoperatively, intraparenchymal hematoma with radiological or clinical signs of the intracranial expansion.
Time Frame: Patients were followed for the duration of hospital stay (average 2 days) and again 2 weeks after the operation.
Population: Complications assessed: Haematoma, Neurological deterioration, Infection
Measure: Number; unit: participants
Groups:
- iMRI: The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a 0.15-T constant magnet is used in all procedures. Subsequently, after the patient's positioning, the preoperative reference examination is routinely carried out (T1+gadolinum, T2 or FLAIR weighted - depending on the pathology, axial 4 mm scans). The entry point, target and optimal biopsy trajectory are then defined by the operator on the basis of the obtained iMRI images. Serial tissue samples (4 from the central and another 4 from the marginal part of the tumour) are collected. Following each operation, a control iMRI (T1-weighted, axial, 4 mm scan examination) is routinely performed to confirm and document the proper targeting and to exclude postoperative hyperacute intraparenchymal bleeding.
  Stereotactic intraoperative magnetic resonance (iMRI)-guided frameless brain tumour biopsy: The PoleStar N20 iMRI system (Medtronic Navigation, Louisville, CO, USA) with a was used in all procedures.
Arm/Group | iMRI | Non-iMRI
Number analyzed (Participants) | 21 | 21
participants | 0 | 1
Statistical Analysis 1: Comparison: iMRI vs Non-iMRI; Test type: Superiority or Other; p = 1.0, Fisher Exact — Fisher's exact test (two-tailed)

2. Primary Outcome: Diagnostic Yield
Description: The diagnostic yield is expressed as the number of patients in whom the histopathological diagnosis was made based of the biological material obtained during the operation.
Time Frame: For each patient 2 weeks after the operation
Measure: Number; unit: participants
Arm/Group | iMRI | Non-iMRI
Number analyzed (Participants) | 21 | 21
participants | 20 | 20
Statistical Analysis 1: Comparison: iMRI vs Non-iMRI; Test type: Superiority or Other; p = 1.0, Fisher Exact

3. Secondary Outcome: Length of Hospital Stay
Description: The preoperative (LOSpre), postoperative (LOSpost) and total length of hospital stay (LOS)
Time Frame: From date of hospitalization until the date of discharge, assessed up to 2 days.
Measure: Median (Full Range); unit: days
Arm/Group | iMRI | Non-iMRI
Number analyzed (Participants) | 21 | 21
days
  Total length of hospital stay | 5 [2 to 13] | 7 [1 to 18]
  The length of preoperative hospital stay | 3 [0 to 8] | 4 [0 to 8]
  The length of postoperative hospital stay | 2 [1 to 6] | 2 [1 to 15]
Statistical Analysis 1: Comparison: iMRI vs Non-iMRI; Total length of hospital stay; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: iMRI vs Non-iMRI; Length of the preoperative hospital stay; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: iMRI vs Non-iMRI; Length of the postoperative hospital stay; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time
Description: the preparation (Tprep), operation (Top) and total operating room (TOR) time
Time Frame: From moment of the transfer to the OR until the moment of transfer out of it, assessed on the day of operation.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | iMRI | Non-iMRI
Number analyzed (Participants) | 21 | 21
minutes
  Total OR time | 111 (24) | 78 (29)
  Time of preparation | 53 (22) | 34 (20)
  Time of the operation | 60 (26) | 44 (20)
Statistical Analysis 1: Comparison: iMRI vs Non-iMRI; Total OR time; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: iMRI vs Non-iMRI; Time of preoperative preparations; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: iMRI vs Non-iMRI; Time of the operation ("skin-to-skin"); Test type: Superiority or Other; p = 0.024, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: A postoperative follow- up head CT was subsequently performed 4 to 6 h after each procedure. All patients were followed up with a clinical examination 2 weeks postoperatively performed by an blinded for the allocation investigator.
Arm/Group | iMRI | Non-iMRI
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No